CLINICAL TRIAL: NCT04064099
Title: Speech Adaptation When Using Mouthguards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Liew (Other)
Responsible Party: Sponsor-Investigator, Amy Liew, Lecturer, Universiti Kebangsaan Malaysia Medical Centre
Organization: Universiti Kebangsaan Malaysia Medical Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UKMPPI/111/8/JEP-2017-439
Record Dates: First submitted 2019-08-07; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Rugby
Keywords: dental trauma; rugby; mouthguard; speech; contact sports
MeSH Terms: conditions — Speech

STUDY DESIGN:
Intervention Model Description: Single group pre- and post- design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rugby Players (Experimental): Rugby player will be given custom-fitted mouthguards to be worn for 6-month
  Interventions: Device: Custom-fitted sports mouthguard

INTERVENTIONS:
Device: Custom-fitted sports mouthguard — Pressure dual laminated technique will be used to fabricate the mouthguards. Ethylene-vinyl acetate (EVA) thermoplastic sheets of 3 mm in thickness with 125 mm diameter (Dentsply International Raintree Essix, Court East Sarasota, USA) will be used. Two 3 mm sheets pressure-laminated together should form an even thickness of 4 mm mouthguard. The design of the mouthguards takes into consideration of the following limits: (i) the labial borders of the mouthguard were extended to within 2 mm of the vestibular reflection, (ii) the palatal margins were trimmed to the cervical area of the palatal surface of the upper teeth, (iii) enclosing the maxillary teeth to the distal surface of the first molars.

SUMMARY:
The aim of this study is to evaluate the speech performance of professional rugby players when using custom-fitted mouthguards over a six-month period. Consented players will be given custom-fitted mouthguards and they will be instructed on the use and care of the mouthguards. At five time points: baseline, immediately following mouthguard use (T1), one-week after- (T2), one-month after- (T3) and six-month after use (T4), participants are required to pronounce four selected phonemes. Three recordings will be made for each phoneme. Spectrspectrographic analysis will be performed to assess the acoustic characteristics of the sound. Concurrently, they will be asked to fill up a questionnaire on self-assessment of oral impairments. Throughout the six-month period, the compliance of wearing mouthguards and the occurrence of dental trauma during training will be monitored on-site by the researcher or if not available, an assigned coach. A 24-hour helpline will be provided as a surveillance tool to monitor problems with mouthguards and dental trauma.

DETAILED DESCRIPTION:
Rugby exposes players to increased risk of dental trauma. Thus, mouthguard use is recommended to provide a resilient surface for shock absorption and impact dissipation. However, some discontinued using mouthguard complaint that general discomfort and speech disturbance are the main barriers to their compliance. The nuisance is largely due to their use of poorly-fitted stock or boil-and-bite mouthguards. Therefore, the primary objective of this study is to evaluate speech adaptations when using custom-fitted mouthguards. The secondary objective is to assess the incidence of dental trauma within the six-month duration of mouthguard use. A prospective study will be carried out at the National Sports Institute. During the first day (T0), a workshop on the prevention and management of dental trauma will be carried out. Then, dental examination, dental impression, and recording of baseline speech performance will be performed. During the second visit (T1), mouthguards delivery, self-assessment of oral impairments, and speech recording will be carried out. After 6-months of monitoring (T2), all participants will be called again to fill in the self-assessment form and final speech performance will be recorded. Data analysis will be carried out to evaluate the self-assessment of speech performance and digital sonography of speech recordings over time. Also, the incidence of dental trauma will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged between 18 and 35;
2. Actively playing rugby;
3. Currently playing in Malaysia Rugby Union;
4. Native speakers of Malay (national language), with the ability to read and write in Malay fluently; and
5. Without any history of either speech or hearing impairment.

Exclusion Criteria:

1. Retired players;
2. National players who did not play rugby within the last six months of the recruitment date; and
3. Players with cleft lip and/or cleft palate; and
4. Players with any history of either speech or hearing impairment.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 35 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Change of speech performance over a six-month period | Baseline (T0), immediately after (T1), one-week after (T2), one-month after (T3) and six-month after (T4) mouthguard use
  Participants will be asked to pronounce the words (paku for phoneme /p/, bola for phoneme /b/, tatu for phoneme /t/, and dadu for phoneme /d/) one by one when it was shown on the computer screen. Three recordings were obtained for each word.

SECONDARY OUTCOMES:
Change of self-assessment of oral impairments over a six-month period | Baseline (T0), immediately after (T1), one-week after (T2), one-month after (T3) and six-month after (T4) mouthguard use
  A questionnaire with a list of oral impairments and five-point Likert scale will be used. The scale name is "Specific problem when using the mouthguard given". Participants will be asked to rate how often they experience the following problems: (i) loose mouthguard, (ii) difficulty speaking, (iii) lisping, (iv) nausea, (v) breathing difficulty, (vi) bulkiness in mouth, (vii) dryness of mouth, (viii) bad breath, (ix) ulcers/sores in mouth, and (x) redness in mouth. The five-point Likert scales have these values: 1=never, 2=rarely, 3=sometimes, 4=often, 5=always. Median score for each question will be reported. Higher values represent worse outcomes.

OTHER OUTCOMES:
Change of self-reported compliance of mouthguard use over a six-month period | Baseline (T0), immediately after (T1), one-week after (T2), one-month after (T3) and six-month after (T4) mouthguard use
  A questionnaire of compliance and five-point Likert scale will be used. The scale name is "Frequency of wearing the mouthguard given". There are two questions: (i) How often do you use the mouthguard during training?, and (ii) How often do you use the mouthguard during competitions? The five-point Likert scales have these values: 1=never, 2=rarely, 3=sometimes, 4=often, 5=always. The median score for each question will be reported. Higher values represent better compliance.
Incidence of dental trauma over a six-month period | Six months, ie. from baseline (T0) to six-month (T3).
  On-site monitoring and 24-hour helpline will be carried out to identify the incidence of dental trauma related to rugby playing. The type of data is count data. The total number of occurrence will be divided by the six months to obtain the incidence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Liew, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mat Zainal MK, Liew AKC, Abdullah D, Soo E, Abdul Hamid B, Ramlee RAM. Changes in oral functions and speech when using custom-fitted mouthguards: An uncontrolled before-and-after study. Dent Traumatol. 2024 Aug;40(4):460-469. doi: 10.1111/edt.12939. Epub 2024 Mar 8. PMID 38459669

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT04064099/Prot_SAP_000.pdf